CLINICAL TRIAL: NCT07242118
Title: Conformal Ablative Radiotherapy in Older Women (CARMEN) With Breast Cancer Undergoing Non-Operative Management
Acronym: CARMEN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Ryan Morse, Assistant Professor, University of Kansas Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2025-CARMEN
Record Dates: First submitted 2025-11-13; First posted 2025-11-21 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer Female
Keywords: Geriatric; ER-positive; HER2-negative

STUDY DESIGN:
Intervention Model Description: Study of women with localized ER+ and HER2- breast cancer receiving non-operative management with SABR delivered to the primary tumor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- SABR Intervention Without Surgery (Single Arm Only) (Experimental): Radiotherapy will be conducted in 5 fractions, every other day. The radiation dose used in this study will use a standard of care post-operative dose of 600 cGy per fraction at 5 total fractions delivered to the clinical target volume. However, since patients in this study will have gross disease and will not have received surgery, a higher dose will be given to the primary tumor itself.
  Study participants may not receive chemotherapeutic agents after enrollment, unless indicated for disease progression. Patients will be allowed to receive CKD 4/6 inhibitors.
  Patients will be allowed on this study whether they do or do not receive anti-hormonal therapy. If a patient has not started endocrine therapy before SABR, ideally, they would initiate endocrine therapy after undergoing SABR. If a patient has already started endocrine therapy before SABR, they may continue during the time of SABR at the discretion of the treating physician, as this is considered safe in this setting.
  Interventions: Radiation: SABR

INTERVENTIONS:
Radiation: SABR — Radiation therapy will consist of either IMRT or 3D CRT. The modality chosen will be based on the plan with the preferable dosimetric variables and determined by the treating radiation oncology physician. SABR will be prescribed to a total dose of 35 Gy to the GTV over the course of 5 fractions (7 Gy per fraction), ideally treated every other day (excluding weekends). The CTV will be prescribed 30 Gy over 5 fractions, ideally treated every other day.

SUMMARY:
This phase II study evaluates SABR as non-operative treatment for women aged 65+ with ER-positive, HER2-negative breast cancer ≤5 cm and no lymph node involvement. Eligible patients, including those previously on endocrine therapy, receive 5 SABR treatments, followed by monitoring of quality of life and assessment of treatment-related toxicity.

DETAILED DESCRIPTION:
This is a prospective, phase II study of women with localized breast cancer receiving non-operative management with SABR delivered to the primary tumor. Patients will be screened that are age 65 and over with invasive breast cancer. Those eligible for the trial will have ER-positive and HER2-negative disease measuring ≤5 cm with negative clinical lymph nodes. Patients that were previously on primary ET, with either stable or progressive disease, will be eligible for this study if other inclusion criteria are met. Participants will receive SABR targeting the tumor consisting of 5 total treatments. Participants will then follow-up as per protocol with quality-of-life assessments and treatment-related toxicity evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent obtained to participate in the study and HIPAA authorization for release of personal health information.
* Women greater than or equal to age 65 years
* Diagnosis of invasive carcinoma of breast undergoing non-operative management
* Previously untreated OR previously treated with primary ET or chemotherapy, with either stable or progressive localized disease.
* Tumor measuring ≤5 cm (cT1-T2) and clinically node negative
* Diagnostic biopsy ER-positive (greater than or equal to 10% ER by immunohistochemistry staining)
* Diagnostic biopsy HER2-negative according to ASCO/CAP guidelines (0 or 1+ following IHC staining or proven negative by in-situ hybridization)
* Suitable for SABR as deemed by the treating radiation oncologist
* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Enrollment in another clinical trial is allowed if there would be no interference with interventions on this trial

Exclusion Criteria:

* Active treatment with systemic chemotherapy for breast cancer. Subjects will need to stop any breast cancer chemotherapy agent before enrollment to be included study.
* Multicentric tumor.
* Clinical or imaging evidence of distant metastases.
* Prior ipsilateral breast or thoracic radiation.
* Autoimmune conditions with associated radiation risks.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — Assigned female at birth
Enrollment: 18 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
1-month post-SABR Physical Well-Being | 1 month
  To estimate the change in the score from baseline to 1-month post-SABR on the BREAST-Q: Physical Well-Being Chest Module in older women receiving non-operative management with SABR for localized breast cancer. Conversion Table will be used to convert the raw scale summed score into a score from 0 (worst) to 100 (best). Higher scores reflect a better outcome.

SECONDARY OUTCOMES:
Patient Reported Outcome | 12 months
  To estimate the change in the score from baseline to 1-month, 6-, and 12-months post-SABR in older women with localized breast cancer undergoing non-operative management using the following BREAST-Q Modules: Satisfaction With Breasts, Adverse Effects of Radiation, Cancer Worry, and Physical-Well Being Chest. Conversion Table will be used to convert the raw scale summed score into a score from 0 (worst) to 100 (best). Higher scores reflect a better outcome.
Treatment Perception | 12 months
  To capture patient perception about treatment with SABR using the three-item survey "Was it worth it?" (WIWI). Scores will be summed from 3 (lowest) to 9 (highest). Higher scores reflect higher satisfaction.
Incidence of SABR-Related Adverse Events [Safety and Tolerability] | 12 months
  To describe treatment-related toxicity at 1-month, 6-, and 12-months post-SABR using Common Terminology Criteria for Adverse Events (CTCAE) in older women with localized breast cancer undergoing non-operative management.
Estimation of Short-term Survival Outcomes | 1 year
  To estimate 1-year progression-free survival (PFS) and overall survival (OS) amongst older women undergoing non-operative management after receiving SABR. Units of Measure include 'alive with disease', 'alive without disease', 'deceased with disease', and 'deceased without disease' at 1-year time interval.

OTHER OUTCOMES:
Exploratory Objective-Estimation of Long-term Survival Outcomes | 2- and 5-years
  To estimate 2-year and 5-year PFS and OS amongst older women undergoing non-operative management after receiving SABR. Units of Measure include qualitative analysis at 2-years and 5-years post-radiation: 'alive with disease', 'alive without disease', 'deceased with disease', and 'deceased without disease'.

CONTACTS AND LOCATIONS:
Overall Officials: Morse, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No